CLINICAL TRIAL: NCT01208584
Title: Brain Function and White Matter Changes in Congenital, Acute and Chronic Spinal Cord Lesions
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Other Study IDs: 306/09
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Paraplegia, Spinal; Myelomeningocele
Keywords: functional MRI,primary motor cortex,spinal cord injury
MeSH Terms: conditions — Paraplegia; Meningomyelocele; Spinal Cord Injuries | interventions — Diffusion Tensor Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Chronic posttraumatic paraplegia: Paraplegic patients (Thoracic level of lesion Th1-Th12), ASIA A, spinal cord injury (SCI) 12-24 months
  Interventions: Other: fMRI, DTI
- Acute posttraumatic paraplegia: Paraplegic patients (Thoracic level of lesion Th1-Th12), ASIA A,SCI 2-6 months,
  Interventions: Other: fMRI, DTI
- Myelomeningocele patients: Myelomeningocele patients (congenital paraplegia, thoracic level of lesion Th1-Th12) ASIA A
  Interventions: Other: fMRI, DTI
- Volunteers: Volunteers without any neurological deficits
  Interventions: Other: fMRI, DTI

INTERVENTIONS:
Other: fMRI, DTI — functional magnetic resonance imaging (fMRI), MR diffusion tensor imaging (DTI)

SUMMARY:
The purpose of this study is to use functional MRI (fMRI) and magnetic resonance (MR) diffusion tensor imaging (DTI) to investigate brain activation and white matter changes in patients with congenital (birth defect of the spinal column), acute and chronic complete spinal cord lesions. The findings of this study may provide a basis to better understand the pathomechanisms underlying the dynamic neurofunctional changes following a spinal cord lesions in man. This understanding is important for the improvement of existing therapies and for the development of new therapeutic approaches.

DETAILED DESCRIPTION:
Recently new approaches to spinal cord repair have been successfully established in animal models. Promising therapies for promoting spinal axonal regeneration in man will be available in the near future. Most research in the field is focussed on the lesion itself and the perilesional spinal cord. The recovery of motor and sensory function is,however, not permitted by local processes at the spinal level only. The whole central nervous system (CNS) reacts to such a condition. Therefore the modulation of motor and sensory function in spinal cord lesioned patients should be reflected in characteristic changes of cortical brain activity, which are accessible to new non-invasive functional neuroimaging techniques such as functional magnetic resonance imaging (fMRI). Changes of white matter due to axonal damage can also be measured qualitatively and quantitatively using MR diffusion tensor imaging (DTI). Those measures may provide a basis to better understand the pathophysiology underlying spinal cord lesions in man, including changes in brain function over time (during rehabilitation) or related to specific treatment. However, there are no studies available yet addressing those topics or providing mechanism-based approaches for determining the time interval of application of novel neuroregenerative drugs. By investigation of brain activation and white matter changes in patients with congenital(myelomeningocele (MMC)), acute and chronic spinal cord lesions (ASIA A) first and fundamental work in this field will be conducted in this study.

ELIGIBILITY:
Inclusion criteria:

* Paraplegic patients (Th1-Th12, ASIA A),
* Myelomeningocele patients (Th1-Th12 ASIA A)
* Acute SCI 2-6 months, chronic SCI 12-24 months

Exclusion criteria:

* Traumatic brain injury (TBI)
* Neurological diseases other than spinal cord lesion
* MRI incompatibility
* Pressure sores
* methicillin-resistant Staphylococcus aureus (MRSA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Paraplegic patients (Thoracic level of lesion Th1-Th12), ASIA A
  * Myelomeningocele patients (congenital paraplegia, thoracic level of lesion Th1-Th12) ASIA A
  * Volunteers without any neurological deficits
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Stippich, Prof, Principal Investigator — University Hospital, Basle - Department of Neuroradiology
Locations (1):
- University Hospital, Basle (only study site!), Basel, Switzerland